CLINICAL TRIAL: NCT03525717
Title: The Effect of Routine vs Late Dinner on Nocturnal Metabolism and Fat Oxidation
Brief Title: Effect of Late Dinner on Nocturnal Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00156120
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: healthy volunteers; metabolism; fat oxidation; obesity; sleep
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Dinner (Active Comparator): Participants will be served dinner and a stable isotope of palmitate to measure fat oxidation, at "routine" dinner time (18:00) followed by a sleep study (23:00). Timing of dinner is the sole intervention distinguishing this arm from late dinner. This arm will cross-over to late dinner in random order.
  Interventions: Dietary Supplement: Routine Dinner; Dietary Supplement: Late dinner
- Late Dinner (Experimental): Participants will be served dinner and a stable isotope of palmitate to measure fat oxidation, at a "late" dinner time (22:00) followed by a sleep study (23:00). Timing of dinner is the sole intervention distinguishing this arm from routine dinner. This arm will cross-over to routine dinner in random order.
  Interventions: Dietary Supplement: Routine Dinner; Dietary Supplement: Late dinner

INTERVENTIONS:
Dietary Supplement: Routine Dinner — Participants will be served dinner at a routine time (18:00), along with with a stable isotope of palmitate to measure fat oxidation overnight.
Dietary Supplement: Late dinner — Participants will be served dinner at a late time (22:00), along with with a stable isotope of palmitate to measure fat oxidation overnight.

SUMMARY:
This study examines the impact of routine dinner time versus late dinner time on nocturnal metabolism. Specifically, investigators will examine plasma profiles of free fatty acids, glucose, insulin, triglycerides, and oxidation of dietary fat.

DETAILED DESCRIPTION:
Obesity is an epidemic contributing to significant global morbidity and mortality. More than simply being a manifestation of excessive eating, obesity and metabolic syndrome may also be the consequence of inappropriate timing of food intake. Specifically, eating more calories later in the day contributes to greater weight gain and metabolic syndrome. The mechanism by which later eating harms metabolism is not fully understood. Meal digestion, absorption, and oxidation can be influenced by circadian rhythm and sleep/wake status. Sleep induces a regulated decrease in metabolic rate, which would be expected to impair the oxidation of ingested fat.

Investigators hypothesize that eating dinner at 10 PM, close to sleep time (11 PM), compared to usual time (6 PM) will lead to impaired nocturnal metabolic profile and reduced fatty acid oxidation of ingested fat. Investigators will test this hypothesis in a randomized crossover study comparing routine dinner (RD) to late dinner (LD) on the nocturnal metabolic profile, and assess oxidation of ingested fat using a stable isotope tracer. If investigators can demonstrate that nocturnal metabolic profile and oxidation of exogenous fat is affected by timing of dinner, investigators can target these pathways for combating obesity and related metabolic consequences.

Study Procedures:

Investigators will perform a randomized cross-over study of RD versus LD on overnight metabolic function in healthy volunteers. Subjects will report to the Bayview Asthma and Allergy center for screening and consent. If participants provide written informed consent, participants will undergo a history and physical examination. Each participant will come to the Clinical Research Unit (CRU) for 2 visits (RD or LD), each comprised of 2 consecutive nights (acclimation night, then study night). The RD and LD visit will be spaced about 3-4 weeks apart, and occur in random order to allow washout of effects and tracer. To account for potential metabolic effects of menstrual cycles, women will studied at the same phase of their menstrual cycle (visits will be ~4 weeks apart). Participants will not have any routine care or current therapy discontinued to enroll in the study.

General visit schedule:

Each of the two visits (3-4 weeks apart) is comprised of two consecutive nights as follows:

* Day 1: Evening admission to the CRU.
* Night 1: Sleep in the CRU without monitoring (acclimation night)
* Day 2: Standardized meals and stable isotope ingestion with either RD or LD, IV sampling (every 60 min)
* Night 2: Sleep in the CRU with Polysomnograph (PSG) and IV sampling (every 60 min)
* Day 3: Standardized breakfast, IV sampling (every 60 min), discharge

Detailed procedures:

Prior to CRU arrival: For 3 days prior to each CRU admission, participants will be asked to keep to a regular sleep-wake cycle, rising at 07:00 h and sleeping at 23:00 and eating 3 meals a day with dinner no later than 19:00.

Day 1 + Night 1: Subjects will undergo a brief history and physical examination. (This can occur on a day remote from admission to the CRU, or on the same afternoon as CRU admission.) At 20:00 subjects will report to the clinical research unit and undergo anthropometric assessment including weight, height, neck, and waist circumference. Participants will be expected to have finished dinner by the time of arrival.

Night 1: Subjects will be provided with a private room in the CRU sleep. Lights will be turned off at 23:00 and turned on at 07:00 the next morning. This is an acclimation night; no polysomnographic monitoring will be performed.

Day 2 + Night 2: Subjects will be awakened at 7:00 AM. Subjects can engage in sedentary activities in the CRU, but participants will not be permitted to sleep or engage in aggressive exercise. Participants will be given four standard meals at 08:00, 13:00, 18:00, and 22:00. The kilocalorie content of each meal, as a percentage of the total daily intake, is shown in the table below and depends on whether participants are under RD or LD conditions

Each meal will have a macronutrient composition of approximately 50% carbohydrate, 30% fat, and 20% protein, but the final diet will be formulated with Institute for Clinical and Translational Research (ICTR) services to reflect typical western diet patterns. Two peripheral IV's will be placed for blood sampling during sleep, with one as a backup in case of failure of one IV. IV tubing will be extended to an adjacent control room so that blood samples can be obtained without disturbing the subject.

Stable Isotope ingestion: Investigators use a validated technique to quantify differences in fatty acid oxidation (FAO) by providing an oral liquid dose of 15 mg/kg body mass of [2H31]palmitate taken with dinner (18:00 on RD night, or 22:00 on LD night). The isotope is dissolved in a warm (60 °C) liquid shake (milk or other emulsifiers) which is provided as a beverage with dinner. FAO will be quantified thereafter by hourly assessment of deuterium incorporation into plasma 2H2O using an isotope ratio MS (IR/MS), eliminating the need for exhaled Carbondioxide (CO2) collection, Variability of Carbondioxide consumption (VCO2) assessment, or acetate correction required with carbon-labeled fatty acid tracers. Subjects will also ingest 0.4 g/kg body mass of H218O so that the total body water volume can be calculated according to the method of Schoeller and van Santen. The FAO rate will be determined by excess plasma 2H times total body water, while percent recovery of deuterium will be determined by dividing by dose of 2H administered.

Night 2: On each study night from 23:00 until 07:00, a PSG will be performed. The sleep study will include electroencephalography, electrooculography, oxygenation, and respiratory effort. Respiratory effort will be measured by thoracoabdominal movement assessed by mercury strain gauges. Surface electrodes will be placed at C3A2 and C3O1, a submental electrode, and left and right electro-oculogram will be used to stage sleep. Electrocardiograph (EKG) tracings will be recorded from three chest electrodes. Continuous measurement of oxygen saturation will be recorded using an ear oximeter (model No 472-1A, Hewlett Packard, Waltham, Mass). Signals from the electroencephalograph, EKG, electromyogram, electrooculogram, respiratory strain gauge, ear oximeter and thermistors will be recorded on a computer with RemLogic software.

Blood work:

Blood samples will be drawn at 60 minute intervals beginning at 5:00 PM and continuing until the next day as shown in fig 1, spanning 20 time points. Each blood sample will be 4 cc in volume and placed into lavender top tubes (EDTA) for centrifugation to obtain plasma. Cells are removed from plasma by centrifugation for 10 minutes at 1500 x using a refrigerated centrifuge. Following centrifugation, plasma will be transferred to cryovials for storage. The morning sample at time of final awakening (7:00 AM) will be 12 cc (3 tubes) since investigators plan additional assays with this sample (lipid panel, inflammatory markers) and 4 cc will be retained as whole blood for future potential analysis. Samples will be frozen at -80°C for research pertaining to metabolic effects of dinner time, with the consent of participants. In total, the blood collected will be approximately 88 cc which is much less than during a blood donation.

Day 3: Participants will be provided with breakfast of similar composition as on day 2, at 08:00. Metabolic response to the meal will be assessed with 4 hourly additional blood samples.

Dual-energy X-ray absorptiometry (DEXA):

A DEXA scan will be used to estimate fat mass, which will be one of the variables analyzed as a predictor of metabolic responses to altered meal time. Only 1 DEXA scan is required per participant and can occur during any of the visit days.

ELIGIBILITY:
Criteria for enrollment and additional information are available at:

https://dinnertimestudy.net/

Inclusion Criteria:

* Healthy male and female adult volunteers, age 18-30.
* Accustomed to a bedtime between 10:00 PM and 1:00 AM.

Exclusion Criteria:

* Sleep disorder including insomnia, sleep apnea, circadian rhythm disorder, restless leg syndrome, narcolepsy, shift work sleep disorder
* Gastroesophageal reflux disease that affects ability to tolerate a dinner close to bed time.
* Chronic use of sedative hypnotics, anxiolytics, opiates
* Use of medications that can affect circadian rhythm (beta blockers, melatonin)
* Active smoking (may interfere with metabolism and CRU activities)
* Diabetes (type 1 or 2)
* Obesity (BMI≥30)
* Pregnant or lactating female (pregnancy test will be required)
* Professional or collegiate athlete

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Free Fatty Acids (FFA, mmol/L) | 2 visits, 4 weeks apart, each visit with 20 time points to assess change over time
  Serial blood samples taken during visit, 20 time points per visit, 2 nights
Glucose (mg/dl) | 2 visits, 4 weeks apart, each visit with 20 time points to assess change over time
  Serial blood samples taken during visit, 20 time points per visit, 2 nights
Insulin (mcU/ml) | 2 visits, 4 weeks apart, each visit with 20 time points to assess change over time
  Serial blood samples taken during visit, 20 time points per visit, 2 nights
Triglycerides (mg/dl) | 2 visits, 4 weeks apart, each visit with 20 time points to assess change over time
  Serial blood samples taken during visit, 20 time points per visit, 2 nights
Oxidation of palmitate (mass spectroscopy) | 2 visits, 4 weeks apart, each visit with 20 time points to assess change over time
  Serial blood samples taken during visit, 20 time points per visit, 2 nights

SECONDARY OUTCOMES:
Polysomnography | 1 sleep study per visit, 4 weeks apart
  Overnight sleep study

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide raw data (without identifying information) to journals or other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be provided upon request within 1 year after publication and will be available to indefinitely.
Access Criteria: The PI will accept requests from other researchers who are examining pertinent outcomes.

REFERENCES:
- [Derived] Gu C, Brereton N, Schweitzer A, Cotter M, Duan D, Borsheim E, Wolfe RR, Pham LV, Polotsky VY, Jun JC. Metabolic Effects of Late Dinner in Healthy Volunteers-A Randomized Crossover Clinical Trial. J Clin Endocrinol Metab. 2020 Aug 1;105(8):2789-802. doi: 10.1210/clinem/dgaa354. PMID 32525525
- See also: Study website — https://dinnertimestudy.net/